CLINICAL TRIAL: NCT04883749
Title: CLL-Frail - A Prospective, Multicenter Phase II Trial of Acalabrutinib in Very Old (≥80y) or Frail CLL-Patients
Brief Title: Efficacy of Acalabrutinib in Very Old or Frail Patients With Treatment-naïve or Relapsed/Refractory CLL
Acronym: CLL-Frail
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL-Frail; 2023-507002-14-00 (EU CTIS Number); 2020-002142-17 (EudraCT Number)
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Chronic Lymphoid Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, B-Cell | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acalabrutinib (Experimental): Acalabrutinib will be administered up to 24 cycles (= approx. 24 months total) until progression of disease (PD) or intolerable toxicity
  Interventions: Biological: Acalabrutinib

INTERVENTIONS:
Biological: Acalabrutinib — Cycle (q28d): Acalabrutinib p.o.100 mg twice daily (BID)
  Other Names: Calquence; ACP-196

SUMMARY:
The aim of this trial is to show the efficacy, safety and feasibility of acalabrutinib in a cohort of CLL-patients ≥80 years or with a FRAIL scale score >2 (5-item questionnaire to be filled out by the patient)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥80 years AND/OR considered too frail for intensive/standard treatment defined by a frailty score of >2 on the FRAIL scale via the patient´s assessment.
2. Have documented CLL requiring treatment according to iwCLL 2018 criteria
3. Ability and willingness to provide written informed consent and to adhere to the study visit schedule and other protocol requirements
4. Glomerular Filtration Rate (GFR) >30ml/min directly measured with 24hr urine collection, calculated according to the modified formula of Cockcroft and Gault (for men: GFR ≈ ((140 - age) x bodyweight)/ (72 x creatinine), for women x 0, 85) or an equally accurate method (Please note: Patients currently on hemodialysis are excluded from participating in the trial)
5. Adequate liver function as indicated by a total bilirubin ≤ 3 x, Aspartate-Aminotransferase/Alanin-Aminotransferase (AST/ ALT) ≤ 3 x the institutional Upper Limit of Normal (ULN) value, unless directly attributable to the patient's CLL or to Gilbert's Syndrome
6. Adequate marrow function independent of growth factor or transfusion support as follows, unless cytopenia is due to marrow involvement of CLL:

   * Absolute neutrophil count ≥ 1.0 × 10^9/L
   * Platelet counts ≥ 30 × 10^9/L; in cases of thrombocytopenia clearly due to marrow involvement of CLL (per the discretion of the investigator); platelet count should be ≥ 10 × 10^9/L if there is bone marrow involvement
   * Total haemoglobin ≥ 9 g/dL (without transfusion support, unless anaemia is due to marrow involvement of CLL)
7. Negative serological testing for hepatitis B (HBsAg negative and anti-HBc negative; patients positive for anti-HBc may be included if PCR for HBV DNA is negative and HBV-DNA Polymerase Chain Reaction (PCR) is performed every month until 12 months after last month of treatment), negative testing for hepatitis C RNA within 6 weeks prior to registration
8. Life expectancy ≥ 3 months
9. Maximum of 1 previous treatment for CLL
10. In case of a recent previous treatment, patients must have recovered from acute toxicities and treatment regimen must be stopped within the following time periods before start of the study treatment in the CLL-Frail trial:

    * chemotherapy ≥ 28 days
    * antibody treatment ≥ 14 days
    * kinase inhibitors (see also exclusion criterion 6), BCL2-antagonists or immunomodulatory agents ≥ 3 days
    * corticosteroids may be applied until the start of the study therapy, these have to be reduced to an equivalent of ≤ 20 mg prednisolone per day during treatment
11. Signed informed consent and, in the investigator's judgment, able to comply with the study protocol

Exclusion Criteria:

1. >1 prior CLL-specific therapy (except corticosteroid treatment administered due to necessary immediate intervention; within the last 14 days before start of study treatment, only dose equivalents up to 20 mg prednisolone are permitted)
2. Transformation of CLL to aggressive Non-Hodgkin's Lymphoma (NHL) e.g. Richter's transformation or prolymphocytic leukaemia
3. Patients with a history of confirmed progressive multifocal leukoencephalopathy (PML)
4. Patients with uncontrolled autoimmune haemolytic anaemia or immune thrombocytopenia
5. Prior exposure to acalabrutinib
6. Progression during previous treatment with another BTK inhibitor, and/or presence of known mutations associated with resistance to therapy, e.g. Bruton´s Tyrosine Kinase (BTK) and Phospholipase C Gamma 2 (PLCg2)
7. Uncontrolled concomitant malignancy, i.e. any concomitant malignancy that may compromise the assessment of CLL stage and the response assessment of the study treatment
8. Eastern Cooperative Oncology Group Performance Status (ECOG) performance status >3
9. Uncontrolled or active infection (including positive SARS-Cov-2 PCR result)
10. Patients with known infection with human immunodeficiency virus (HIV)
11. Significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 3 months of screening, or any class 4 cardiac disease as defined by the New York Heart Association Functional Classification at Screening (Please note: Subjects with controlled, asymptomatic atrial fibrillation are allowed to enroll on study)
12. Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening
13. Significantly increased risk of bleeding according to the investigator´s evaluation, e.g. due known bleeding diathesis (e.g. von-Willebrandt´s disease or hemophilia), major surgical procedure ≤ 4 weeks or stroke/intracranial hemorrhage ≤ 6 months
14. Use of investigational agents which might interfere with the study drug within 28 days prior to registration for study screening
15. Requirement of therapy with strong CYP3A4 inhibitors/inducers or anticoagulant with phenprocoumon (marcumar) or other vitamin K-antagonists (Please note: Switch to alternative anticoagulants for vitamin K antagonists is permitted)
16. Inability to swallow tablets
17. Legal incapacity
18. Prisoners or subjects who are institutionalized by regulatory or court order
19. Persons who are in dependence to the sponsor or an investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) at initial response assessment | At initial response assessment (approx. 6 months after initiation of therapy)
  Proportion of patients having achieved complete response (CR), complete response with incomplete bone marrow recovery (CRi) or partial response (PR) as response (according to the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 guidelines)

SECONDARY OUTCOMES:
ORR at final restaging | At final restaging (approx. 24 months after initiation of therapy)
  Proportion of patients having achieved complete response (CR), complete response with incomplete bone marrow recovery (CRi) or partial response (PR) as response (according to the iwCLL 2018 guidelines)
Overall survival (OS) | Up to 24 month
  Time from the date of registration to the date of death due to any cause
Progression-free survival (PFS) | Up to 24 month
  Time from the date of registration to the date of first occurrence of disease progression or relapse (according to iwCLL 2018 criteria) or death from any cause, whichever occurs first
Event-free survival (EFS) | Up to 24 month
  Time from the date of registration to the first occurrence of progression or relapse (according to iwCLL 2018 criteria), death from any cause or initiation of a subsequent anti-leukemic treatment, whichever occurs first
Time to next CLL treatment (TTNT). | Up to 24 month
  Time from date of registration to the date of initiation of subsequent anti-leukemic treatment
Safety parameters: Adverse events (AE) and adverse events of special interest (AESI) | Up to 24 month
  Type, frequency, and severity of AEs and AESIs

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Eichhorst, Prof., Principal Investigator — Department I of Internal Medicine, University Hospital Cologne
Locations (20):
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck
  - Hanusch Krankenhaus, Vienna
- Germany (18):
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Universitätsklinik Köln, Cologne
  - Donau-Isar-Klinikum Deggendorf Hämatologie/Onkologie, Deggendorf
  - Oncoresearch Institut für klinische Studien GbR, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Onkologische Kooperation Harz, Goslar
  - OncoResearch Lerchenfeld, Hamburg
  - MediProjekt GBR, Hanover
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Praxis fuer Haematologie und Onkologie, Koblenz
  - H.O.T Praxis Landshut, Landshut
  - Lübecker Onkologische Schwerpunktpraxis, Lübeck
  - Gemeinschaftspraxis Haematologie und Onkologie, Magdeburg
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Ravensburg
  - Universitaetsklinikum Ulm, Ulm
  - Hämatologisch Onkologische Schwerpunktpraxis, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simon F, Ligtvoet R, Bohn JP, Nosslinger T, von Tresckow J, Liersch R, Gaska T, Jentsch-Ullrich K, Gartner M, Wolff T, Schwaner I, Wolf D, Schneider C, Vehling-Kaiser U, Ritgen M, Spoer C, Eckart M, Decker T, Chakupurakal G, Schottker B, Kisro J, Kreuzer KA, Tausch E, Stilgenbauer S, Robrecht S, Stumpf J, Fink AM, Furstenau M, Fischer K, Goede V, Hallek M, Eichhorst B. Acalabrutinib treatment for older (aged >/=80 years) and/or frail patients with CLL: primary end point analysis of the CLL-Frail trial. Blood. 2025 Dec 25;146(26):3153-3162. doi: 10.1182/blood.2025028550. PMID 40906922
- See also: Click here for more information about this study: CLL-Frail (German CLL Study Group) — https://www.dcllsg.com/cll-frail/